CLINICAL TRIAL: NCT03476824
Title: PelvFx - Pelvic Fractures in the Elderly Patient Influence of Fracture Classification According to Rommens & Hofmann on Mobility, Operation and Independence
Brief Title: Pelvic Fractures in the Elderly
Acronym: PelvFx
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-01859; ch18Ramser
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Pelvic Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the project is to predict the patient under conservative therapy as a function of the patient Classification of Rommens and Hofmann and other potential prognostic factors. A corresponding prognostic score may be used in the future by patients and attending physicians support joint decision between surgical and conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pelvic fracture after low-energy trauma
* Treatment in the years 2006 to 2016
* patients equal to or older than 60 years

Exclusion Criteria:

* Pelvic fracture after a high-energy space
* Pathological fracture in the area of a tumor or a bony metastasis
* Existence of a documented refusal

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients are filtered out of our electronic patient system on the basis of the diagnosis "pelvic ring fracture". Subsequently, patients under the age of 60 and patients after high-energy trauma are excluded.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
mortality | from pelvic fracture until year 1
  number of patients who died within one year after pelvic fracture
loss of independence | from pelvic fracture until year 1
  loss of independence defined as number of patients leaving their own home and starting to live in a retirement home or asylum within one year after pelvic fracture

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Ramser, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Switzerland, Traumatology, Basel, Switzerland